CLINICAL TRIAL: NCT01922063
Title: Long Term Follow-up of Comprehensive Physiotherapy Following Disc Herniation Operation: Results of a Randomized Clinical Trial
Brief Title: Physiotherapy Following Disc Surgery: Long Term Follow-up of a RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Gerold Ebenbichler, Prof Dr Gerold Ebenbichler, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMR_Ebe01/2009; EK Nr. 301/2009 (Other: Ethics committee, Medical University of Vienna)
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Intervertebral Disc Displacement
Keywords: disc herniation surgery; physiotherapy, exercise therapy; randomized; long term; follow up
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Physiotherapy Intervention (Experimental): 20 treatment sessions of a comprehensive physiotherapy program, 12 weeks' duration, with custom tailored instructions by the supervising physician; physicians discussed the course of therapy with the physiotherapist 1x/week. Patients had been treated by physiotherapist according to written prescriptions. Duration of treatment 30 min/ session. Patients were encouraged to practice regular home exercise.
  Interventions: Behavioral: Physiotherapy Intervention
- Sham neck massage (Sham Comparator): received twenty sessions "sham" neck massage of 30 minutes' duration each with the patients lying in supine position on a massage bed and the head of the patient resting on the therapist's knees
  Interventions: Behavioral: Sham neck massage
- No therapy (No Intervention): no further therapy, patients were asked to "wait and see" for the first three months after operation, and no particular treatment was planned

INTERVENTIONS:
Behavioral: Physiotherapy Intervention — 20x 30 min sessions of physiotherapy
  Arms: Physiotherapy Intervention
Behavioral: Sham neck massage — 20x 30 minutes sessions of neck massage
  Arms: Sham neck massage

SUMMARY:
Hitherto no comprehensive long-term follow-up data of 10 years and more have been obtained from survivors of disc surgery that would have considered the type of postoperative care.

Objectives: 1) To evaluate the long-term effects of postoperative comprehensive physiotherapy starting 1 week after lumbar disc surgery. 2) To assess the relative risk of segmental instability in the operated segment 12 years following lumbar disc surgery.

DETAILED DESCRIPTION:
Design: Twelve years' follow-up of a three-armed, randomized, controlled, single blinded clinical trial. Setting: Outpatient department of Physical Medicine & Rehabilitation. Participants: Of 120 patients following first-time, uncomplicated lumbar disc surgery who participated in the original study are invited to a 12 years follow-up examination. Interventions: In the original study, patients had been randomly assigned to "comprehensive physiotherapy", "sham intervention" (neck massage), or no therapy. Measurements: Low Back Pain Rating Score (LBPRS; Manniche 1993), functional X-rays of the lumbar spine. All data are collected by blinded students and physicians at the Department of PM&R, Vienna Medical University.

ELIGIBILITY:
Inclusion Criteria:

* all patients who had undergone a first time uncomplicated disc surgery for lumbar vertebral disc herniation who had taken part in the original RCT and had completed the treatment originally allocated
* all patients who had undergone a first time uncomplicated disc surgery for lumbar vertebral disc herniation who had taken part in the original RCT and had not completed the treatment originally allocated

Exclusion Criteria:

* n.a.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 1996-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Low back pain rating scale (LBP-RS) | 12 years after Randomization
  The LBP-RS measures the health concepts of pain, disability, and physical impairment. Both the original and the translated version of the LBP rating scale are highly reliable within and between raters, uni-dimensional and are shown to have satisfactory construct validity. The sum score ranges from 130 (worst) to 0 (best) and is the composite of 3 subscores (pain, disability, and physical function).

SECONDARY OUTCOMES:
Satisfaction with treatment | 12 years
  Ratings on a 5-point Likert scale (1= completely recovered to 5= dramatically worse as compared to baseline
Use of health care resources | 12 years
  questions related to the use of health care resources because of back pain, and the necessity of reoperation of a disc herniation
Psychological questionnaires | 12 years
  Fear Avoidance beliefs questionnaire, MOS 36-Item Short Form Health Survey, Heidelberger Pain Inventory Symptom Checklist-90R (SCL-90R) Beck Depression Inventory (BDI)

OTHER OUTCOMES:
X Rays | 12 years
  Functional X rays of the lumbar spine

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Ebenbichler, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Dept Physical Medicine & Rehabilitation, MUV, AKH, Vienna, Austria